CLINICAL TRIAL: NCT06618040
Title: Bedtime Stories: Tailored Sleep Health Messaging for Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Judith Owens, Professor of Neurology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00047237
Record Dates: First submitted 2024-08-14; First posted 2024-10-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Sleep; Health-Related Behavior
MeSH Terms: conditions — Health Behavior | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Health Education Program for Caregivers (Experimental): The BTS-C is an online sleep health education program that is located on a mobile application. The BTS-C utilizes asynchronous avatar-based interactive learning and educational content and videos that are tailored to the caregivers' goals and expectations, paired with targeting messages for change surrounding principles of sleep health practices. The modules will be completed over the course of 6 weeks.
  Interventions: Behavioral: Bedtime Stories Sleep Health Education Program for Caregivers (BTS-C)

INTERVENTIONS:
Behavioral: Bedtime Stories Sleep Health Education Program for Caregivers (BTS-C) — The BTS-C includes 6 educational modules on different topics related to sleep health: principles of healthy sleep practices include sleep routines, the sleep environment, considerations for screen time, timing of sleep and activities surrounding sleep, expectations for healthy sleep and sleep duration. Caregivers will also receive a combination of tailored messages or prompts to explore progress, identify strategies for change, and goal setting.

SUMMARY:
To date, there are very few established sleep health education models targeting caregivers of school-aged children from historically marginalized and/or low income communities. To address this significant gap, this project seeks to examine the feasibility, acceptability, and usability of the Bedtime Stories Sleep Health Education Program to improve sleep behavior. Bedtime Stories is a multi-stakeholder (health care providers, school-aged children, and caregivers of school-aged children) and a multi-component program. The caregiver component of the program utilizes mobile health technology with targeted and tailored sleep health messaging for caregivers of school-aged children. Addressing these aims will help to mitigate gaps in the delivery of health care services to caregivers and families in low income and historically marginalized communities, where services and interventions are scant.

DETAILED DESCRIPTION:
Healthy sleep practices are a fundamental component of sleep education interventions designed to prevent sleep problems from developing (Masten et al., 2006) and aide in managing existing sleep disorders such as insomnia in children (Moore et al., 2007). Although poor sleep is linked to a host of negative outcomes, sleep health may also be viewed in a positive light, i.e., "sleep wellness" that places the emphasis on the benefits of good sleep and its importance to overall health maintenance and improvement. Indeed, both the positive and negative aspects of sleep are highly relevant with regards to developing sleep health educational programs, while providing concrete targets for health promotion, wellness and prevention. Fostering healthy sleep habits in children and adolescents builds the foundation for healthy sleep habits in adulthood (Galland et al., 2010). A major challenge to identifying sleep concerns in children is that identification often relies on parent reported concerns, professional clinical judgment, and the presence of symptomatology that changes with age. The early diagnosis of sleep concerns is a key factor to enable access to interventions that improve sleep health. To address this critical gap requires targeted interventions tailored to healthcare providers, particularly those serving communities and populations most in need.

Interventions for caregivers focused on sleep health, including sleep health practice, building and supporting routines, and consistent sleep schedules are integral features to sleep. Settings to promote healthy sleep practices including well-child visits. The well-child visit is an opportunity to educate parents about normal sleep in children and provide strategies to prevent sleep problems from either developing, or if problems already exist from becoming chronic. Community health centers which serve both children and adults, afford unique opportunities to incorporate screening and the prevention of sleep disorders; and deliver coordinated health messages to parents and children in order to effect positive behavioral change within the entire family.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* Caregivers of school-aged children (5-11 years of age) that receive care at participating community healthcare centers in the Boston area
* English fluency

Exclusion Criteria:

* Planning on moving within the next 3 months
* Does not live in the home with the child

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Knowledge, Perceptions, and Practices | Follow Up, after 8 weeks
  Using the parent Knowledge, Attitudes, Self-Efficacy, and Beliefs scale (adapted questionnaire), 19-item questionnaire; minimum score is 19 and maximum score is 95. A higher score means better sleep habits.
Feasibility, acceptability, and usability | Follow Up, after 8 weeks
  Using the Brief Feedback questionnaire (BFQ), 15-item questionnaire; total score
Assessment of Child Sleep | 1 week baseline, 1 week follow up, entire study
  Using a sleep diary (1-week; sleep duration, total sleep time) and the Fitbit Inspire 3 (sleep duration, sleep efficiency, regulatory of sleep time)
Child Sleep Health | Baseline (at week 0), Follow Up (after 8 weeks)
  Using the Child Sleep Habits Questionnaire: 22-item parent report; Bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep disordered breathing, daytime sleepiness; total score

SECONDARY OUTCOMES:
Child Sleep Environment | Baseline (at week 0)
  Using the Children's Adolescents' Sleep Environment Scale (CASES): 13-item parent report; total score
Child Sleep Disturbance Impairments | Baseline (at week 0), Follow Up (after 8 weeks)
  Using the PROMIS: 8-item parent report, total score; and the disturbance 8-item parent report, total score; impairment
Assessment of parent/caregiver sleep | Baseline (at week 0), Follow Up (after 8 weeks), Entire Study (8 weeks)
  Using the Pittsburgh Sleep Quality Index (PSQI), 19-item questionnaire: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleeping medication, daytime dysfunction, total score; and the Fitbit Inspire 3: Baseline and follow up; sleep duration, sleep efficiency, regulatory of sleep time
Caregiver Stress | Baseline (at week 0), Follow Up (after 8 weeks)
  Using the Parent Stress Index-Short Form (PSI), 36-item questionnaire: parent distress, parent-child dysfunctional interaction, difficult child; total score

CONTACTS AND LOCATIONS:
Overall Officials: Judith Owens, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mindell JA, Bartle A, Wahab NA, Ahn Y, Ramamurthy MB, Huong HT, Kohyama J, Ruangdaraganon N, Sekartini R, Teng A, Goh DY. Sleep education in medical school curriculum: a glimpse across countries. Sleep Med. 2011 Oct;12(9):928-31. doi: 10.1016/j.sleep.2011.07.001. Epub 2011 Sep 16. PMID 21924951
- [Background] Owens JA, Jones C. Parental knowledge of healthy sleep in young children: results of a primary care clinic survey. J Dev Behav Pediatr. 2011 Jul-Aug;32(6):447-53. doi: 10.1097/DBP.0b013e31821bd20b. PMID 21546852